CLINICAL TRIAL: NCT05956899
Title: A Comparison Between Palonosetron And Ondansetron As Prophylaxis Against Postoperative Nausea and Vomiting In Idiopathic Scoliosis Surgery: A Randomised Trial
Brief Title: Palonosetron vs Ondansetron In PONV Prophylaxis Among Idiopathic Scoliosis Patients
Acronym: PONV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Dr. Siti Nadzrah Yunus, Doctor, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20221016-11624
Record Dates: First submitted 2023-05-21; First posted 2023-07-24 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Idiopathic Scoliosis; Postoperative Nausea and Vomiting
Keywords: Antiemetics; Dexamethasone; Ondansetron; Palonosetron; Scoliosis; PONV
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Scoliosis | interventions — Palonosetron; Ondansetron

STUDY DESIGN:
Intervention Model Description: After taking informed consent and recruitment of eligible participants, they will be randomized using a sequentially numbered, opaque sealed envelope (SNOSE) method. 74 radio-opaque envelopes will be prepared according to two groups: 37 participants for each Group A, Palonosetron and Group B, Ondansetron. Group A will receive IV palonosetron 1.5mcg/kg prior to commencement of general anaesthesia; while Group B will receive IV ondansetron 0.15mg/kg at the start of wound closure.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): Group A will receive a stat dose of IV palonosetron 1.5mcg/kg prior to commencement of general anaesthesia.
  Interventions: Drug: Palonosetron
- Group B (Active Comparator): Group B will receive a stat dose of IV ondansetron 0.15mg/kg at the start of wound closure.
  Interventions: Drug: Ondansetron

INTERVENTIONS:
Drug: Palonosetron — IV palonosetron 1.5mcg/kg prior to commencement of general anaesthesia
  Arms: Group A
Drug: Ondansetron — IV ondansetron 0.15mg/kg at the start of wound closure
  Arms: Group B

SUMMARY:
The goal of this clinical trial is to compare the effectiveness of two antiemetic drugs, palonosetron and ondansetron, when given alongside dexamethasone as a preventive measure against early and delayed postoperative nausea and vomiting (PONV) in adult and adolescent patients with idiopathic scoliosis undergoing posterior spinal fusion surgery under total intravenous anesthesia (TIVA).

The main questions the study aims to answer are:

* How effective is palonosetron compared to ondansetron, both combined with dexamethasone, in preventing PONV after scoliosis surgery?
* Are there any differences in the need for rescue antiemetics, occurrence of adverse effects related to the study drugs, and patient satisfaction between the two treatment groups?

Participants in the study will be randomly assigned to receive either palonosetron or ondansetron in addition to dexamethasone as part of their anesthesia and antiemetic regimen. The incidence and/ or severity of nausea, vomiting and retching will be assessed at 1 hour, 4 hours, 12 hours, 24 hours and 48 hours after surgery.

DETAILED DESCRIPTION:
BACKGROUND/ JUSTIFICATION Postoperative nausea and vomiting (PONV) is a common complication following surgery and can cause significant morbidity. It occurs in 20-30% of the general population and up to 75-80% in high-risk groups. Children have a higher incidence of PONV compared to adults. PONV can occur at various timeframes after surgery and has clinical and financial consequences, including wound complications, dehydration, and prolonged hospitalization. Prevention and treatment of PONV are crucial for comprehensive perioperative care.

Posterior spinal fusion surgery for idiopathic scoliosis is a complex and painful procedure, increasing the risk of PONV. Various strategies can be employed to mitigate these risks, such as adequate hydration, the use of intravenous antiemetics, avoiding volatile anesthetics, and adopting a multimodal analgesic approach. Dexamethasone and anti-serotonergic drugs like ondansetron are commonly used antiemetics due to their efficacy and safety profiles. Dexamethasone is particularly favored for its long duration of action and pain-reducing effects.

Palonosetron, a second-generation anti-serotonergic drug, has a unique pharmacokinetic profile with a prolonged duration of action. It may be more beneficial for patients on prolonged opioid-based analgesic regimens. However, its higher cost and inconsistent study findings limit its widespread use, especially in scoliosis patients undergoing spinal fusion surgery.

Total intravenous anesthesia (TIVA) is recommended for high-risk PONV patients, as it reduces the emetogenic effect of volatile anesthetics. Propofol, used in TIVA, is itself an effective antiemetic. TIVA with propofol has been shown to be as effective as giving a single antiemetic and can further reduce the risk of PONV when combined with other prophylactic antiemetics.

The standard practice for managing PONV involves the administration of two antiemetics and considering TIVA for high-risk patients. This study aims to compare the effectiveness of palonosetron and ondansetron when administered alongside dexamethasone in scoliosis patients undergoing spinal fusion under TIVA. The study will also evaluate the number of rescue antiemetics needed, assess adverse effects, and measure patient satisfaction.

The study will be randomized and double-blinded, to be conducted in Universiti Malaya Medical Centre (UMMC). The sample size is calculated to be 92 participants, after taking into account a 20% dropout rate. Adult and adolescent idiopathic scoliosis patients undergoing posterior spinal fusion surgery will be eligible for the study. Written informed consent will be obtained from participants or their guardians, and assent will be obtained from adolescent participants. Patients will be randomized to receive either palonosetron or ondansetron along with dexamethasone.

The study will follow standard anesthetic techniques, including TIVA with remifentanil and propofol. Intravenous injections of the study drugs or placebo will be given during surgery, and dexamethasone will be administered as a baseline antiemetic. Morphine will be administered before the end of surgery for pain management.

ELIGIBILITY:
Inclusion Criteria:

* Age of 10 years and above
* American Society of Anaesthesiologists (ASA) I-II Physical Status

Exclusion Criteria:

* History of allergy to serotonin receptor antagonists or dexamethasone
* Obesity with a body mass index (BMI) of 34 and above
* Body weight of less than 30kg
* Active smoker
* History of gastroesophageal reflux disease/ other gastrointestinal diseases associated with vomiting
* History of motion sickness
* History of nausea or vomiting within 24 hours before the surgery
* Administration of antiemetics/ steroids/ psychoactive medications within 24 hours before the surgery
* Require mechanical ventilation postoperatively
* History of cardiac arrhythmias
* Prolonged QT (QTc is prolonged if > 440ms in men or > 460ms in women

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-05-02 (Actual)

PRIMARY OUTCOMES:
Incidence of PONV | At 1 hour after surgery
  To compare the effectiveness of palonosetron and ondansetron when administered alongside dexamethasone as prophylaxis against early and delayed postoperative nausea and vomiting (PONV) in adult and adolescent idiopathic scoliosis patients undergoing posterior spinal fusion surgery under total intravenous anaesthesia.
Incidence of PONV | At 4 hours after surgery
  To compare the effectiveness of palonosetron and ondansetron when administered alongside dexamethasone as prophylaxis against early and delayed postoperative nausea and vomiting (PONV) in adult and adolescent idiopathic scoliosis patients undergoing posterior spinal fusion surgery under total intravenous anaesthesia.
Incidence of PONV | At 12 hours after surgery
  To compare the effectiveness of palonosetron and ondansetron when administered alongside dexamethasone as prophylaxis against early and delayed postoperative nausea and vomiting (PONV) in adult and adolescent idiopathic scoliosis patients undergoing posterior spinal fusion surgery under total intravenous anaesthesia.
Incidence of PONV | At 24 hours after surgery
  To compare the effectiveness of palonosetron and ondansetron when administered alongside dexamethasone as prophylaxis against early and delayed postoperative nausea and vomiting (PONV) in adult and adolescent idiopathic scoliosis patients undergoing posterior spinal fusion surgery under total intravenous anaesthesia.
Incidence of PONV | At 48 hours after surgery
  To compare the effectiveness of palonosetron and ondansetron when administered alongside dexamethasone as prophylaxis against early and delayed postoperative nausea and vomiting (PONV) in adult and adolescent idiopathic scoliosis patients undergoing posterior spinal fusion surgery under total intravenous anaesthesia.

SECONDARY OUTCOMES:
Number of Participants Developing Postoperative Nausea Vomiting Requiring Rescue Antiemetic Within 48 hours After Surgery | At 1 hour, 4 hours, 12 hours, 24 hours and 48 hours after surgery
  Any occurrence of severe nausea and retching with visual analogue scale score ≥4; and vomiting of 1 or more episodes will be treated with the rescue drug IV metoclopramide. For adolescent subjects (aged less than 18 years old), IV metoclopramide will be given at 0.2mg/kg, with a maximum dose of 10 mg intravenously up to 3 times per day. For adult patients (18 years old and above), IV metoclopramide 10mg will be given, up to 3 times per day. If there is any further occurrence of PONV within 8 hours of administration of IV metoclopramide, a second line of rescue antiemetic, IV ondansetron 4mg, will be administered to participants in both arms of the study. The administration of any rescue medications will be recorded and taken into account during data processing.
Number of Participants Developing Adverse Effects Related to the Study Drugs. | Overall, assessed at 48 hours after surgery
  Such as headache, dizziness and constipation
Degree of patient satisfaction as represented on the Visual Analogue Scale | Overall, assessed at 48 hours after surgery
  On a scale of 1 (least satisfied) to 5 (most satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Siti Nadzrah Binti Yunus, MAnaes, MBBS, Principal Investigator — Universiti Malaya
Locations (1):
- University Malaya, Pantai Valley, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kumar A, Solanki SL, Gangakhedkar GR, Shylasree TS, Sharma KS. Comparison of palonosetron and dexamethasone with ondansetron and dexamethasone for postoperative nausea and vomiting in postchemotherapy ovarian cancer surgeries requiring opioid-based patient-controlled analgesia: A randomised, double-blind, active controlled study. Indian J Anaesth. 2018 Oct;62(10):773-779. doi: 10.4103/ija.IJA_437_18. PMID 30443060
- [Background] Kotiniemi LH, Ryhanen PT, Valanne J, Jokela R, Mustonen A, Poukkula E. Postoperative symptoms at home following day-case surgery in children: a multicentre survey of 551 children. Anaesthesia. 1997 Oct;52(10):963-9. doi: 10.1111/j.1365-2044.1997.203-az0338.x. PMID 9370838
- [Background] Villeret I, Laffon M, Duchalais A, Blond MH, Lecuyer AI, Mercier C. Incidence of postoperative nausea and vomiting in paediatric ambulatory surgery. Paediatr Anaesth. 2002 Oct;12(8):712-7. doi: 10.1046/j.1460-9592.2002.00952.x. PMID 12472709
- [Background] Patel RI, Hannallah RS. Anesthetic complications following pediatric ambulatory surgery: a 3-yr study. Anesthesiology. 1988 Dec;69(6):1009-12. doi: 10.1097/00000542-198812000-00044. No abstract available. PMID 3195743
- [Background] Rowley MP, Brown TC. Postoperative vomiting in children. Anaesth Intensive Care. 1982 Nov;10(4):309-13. doi: 10.1177/0310057X8201000402. PMID 7158749
- [Background] Awad IT, Moore M, Rushe C, Elburki A, O'Brien K, Warde D. Unplanned hospital admission in children undergoing day-case surgery. Eur J Anaesthesiol. 2004 May;21(5):379-83. doi: 10.1017/s0265021504005058. PMID 15141796
- [Background] Kovac AL. Update on the management of postoperative nausea and vomiting. Drugs. 2013 Sep;73(14):1525-47. doi: 10.1007/s40265-013-0110-7. PMID 24057415
- [Background] Dolin SJ, Cashman JN, Bland JM. Effectiveness of acute postoperative pain management: I. Evidence from published data. Br J Anaesth. 2002 Sep;89(3):409-23. PMID 12402719
- [Background] Golembiewski J, Chernin E, Chopra T. Prevention and treatment of postoperative nausea and vomiting. Am J Health Syst Pharm. 2005 Jun 15;62(12):1247-60; quiz 1261-2. doi: 10.1093/ajhp/62.12.1247. PMID 15947124
- [Background] Kovac AL. Prevention and treatment of postoperative nausea and vomiting. Drugs. 2000 Feb;59(2):213-43. doi: 10.2165/00003495-200059020-00005. PMID 10730546
- [Background] Apfel CC, Laara E, Koivuranta M, Greim CA, Roewer N. A simplified risk score for predicting postoperative nausea and vomiting: conclusions from cross-validations between two centers. Anesthesiology. 1999 Sep;91(3):693-700. doi: 10.1097/00000542-199909000-00022. PMID 10485781
- [Background] Apfel CC, Kranke P, Eberhart LH, Roos A, Roewer N. Comparison of predictive models for postoperative nausea and vomiting. Br J Anaesth. 2002 Feb;88(2):234-40. doi: 10.1093/bja/88.2.234. PMID 11883387
- [Background] Gan TJ, Belani KG, Bergese S, Chung F, Diemunsch P, Habib AS, Jin Z, Kovac AL, Meyer TA, Urman RD, Apfel CC, Ayad S, Beagley L, Candiotti K, Englesakis M, Hedrick TL, Kranke P, Lee S, Lipman D, Minkowitz HS, Morton J, Philip BK. Fourth Consensus Guidelines for the Management of Postoperative Nausea and Vomiting. Anesth Analg. 2020 Aug;131(2):411-448. doi: 10.1213/ANE.0000000000004833. PMID 32467512
- [Background] Eberhart LHJ, Geldner G, Kranke P, Morin AM, Schauffelen A, Treiber H, Wulf H. The development and validation of a risk score to predict the probability of postoperative vomiting in pediatric patients. Anesth Analg. 2004 Dec;99(6):1630-1637. doi: 10.1213/01.ANE.0000135639.57715.6C. PMID 15562045
- [Background] Palmer GM, Pirakalathanan P, Skinner AV. A multi-centre multi-national survey of anaesthetists regarding the range of anaesthetic and surgical practices for paediatric scoliosis surgery. Anaesth Intensive Care. 2010 Nov;38(6):1077-84. doi: 10.1177/0310057X1003800619. PMID 21226441
- [Background] Ho CM, Wu HL, Ho ST, Wang JJ. Dexamethasone prevents postoperative nausea and vomiting: benefit versus risk. Acta Anaesthesiol Taiwan. 2011 Sep;49(3):100-4. doi: 10.1016/j.aat.2011.06.002. PMID 21982171
- [Background] Wakamiya R, Seki H, Ideno S, Ihara N, Minoshima R, Watanabe K, Sato Y, Morisaki H. Effects of prophylactic dexamethasone on postoperative nausea and vomiting in scoliosis correction surgery: a double-blind, randomized, placebo-controlled clinical trial. Sci Rep. 2019 Feb 14;9(1):2119. doi: 10.1038/s41598-019-38764-8. PMID 30765809
- [Background] Kloth DD. New pharmacologic findings for the treatment of PONV and PDNV. Am J Health Syst Pharm. 2009 Jan 1;66(1 Suppl 1):S11-8. doi: 10.2146/ashp080462. PMID 19106333